CLINICAL TRIAL: NCT02047734
Title: A Phase 2/3, Multi-center, Randomized, Double-blind, Placebo-controlled (Part A) and Double-blind, Double-dummy, Active-controlled (Part B), Parallel Group Study to Evaluate the Efficacy and Safety of RPC1063 Administered Orally to Relapsing Multiple Sclerosis Patients
Brief Title: Efficacy and Safety Study of Ozanimod in Relapsing Multiple Sclerosis
Acronym: RADIANCE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RPC01-201-PartB; 2012-002714-40 (EudraCT Number)
Record Dates: First submitted 2014-01-26; First posted 2014-01-28 (Estimated); Results first posted 2021-02-11 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-01

CONDITIONS: Relapsing Multiple Sclerosis
MeSH Terms: interventions — ozanimod; Interferon beta-1a

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Ozanimod 0.5 mg (Experimental): Ozanimod 0.5 mg oral capsules daily and a weekly intramuscular placebo injection (identical in appearance to Interferon) for 24 months.
  Interventions: Drug: Ozanimod; Drug: Interferon beta-1a placebo
- Ozanimod1 mg (Experimental): Ozanimod 1 mg oral capsules daily and a weekly intramuscular placebo injection (identical in appearance to Interferon) for 24 months.
  Interventions: Drug: Ozanimod; Drug: Interferon beta-1a placebo
- Interferon β-1a (Active Comparator): interferon beta-1a (IFN β-1a) 30 µg intramuscular (IM) injection weekly and matching placebo capsules (identical in physical appearance to ozanimod) orally daily for 24 months.
  Interventions: Drug: Ozanimod placebo; Drug: Interferon beta-1a

INTERVENTIONS:
Drug: Ozanimod — Oral capsule, daily for 24 months
  Other Names: RPC1063; Zeposia®
  Arms: Ozanimod 0.5 mg; Ozanimod1 mg
Drug: Ozanimod placebo — Oral capsule, daily for 24 months
  Arms: Interferon β-1a
Drug: Interferon beta-1a — Intramuscular injection, 30 µg, weekly for 24 months
  Other Names: Avonex
  Arms: Interferon β-1a
Drug: Interferon beta-1a placebo — Intramuscular injection, weekly for 24 months
  Arms: Ozanimod 0.5 mg; Ozanimod1 mg

SUMMARY:
This study is a two-part trial consisting of Part A (see NCT01628393) and Part B, presented within this record.

The primary objective of Part B is to assess whether the clinical efficacy of ozanimod (RPC1063) is superior to interferon beta-1a (IFN β-1a; Avonex®) in reducing the rate of clinical relapses at the end of Month 24 in patients with relapsing multiple sclerosis (RMS).

DETAILED DESCRIPTION:
This clinical trial (RPC01-201; RADIANCE) consisted of 2 parts, each reported separately on ClinicalTrials.gov: Part A (NCT01628393) and Part B (this record).

Part A was a phase 2 study in which two doses of ozanimod were administered daily for 24 weeks with an efficacy and safety comparison to a placebo control and is reported separately as ClinicalTrials.gov record NCT01628393.

Part B, reported herein, was a phase 3 study in which two doses of ozanimod were administered daily for a 24 month period compared to an active control, interferon β-1a. Participants were allowed to enroll in the open-label extension study RPC01-3001 (NCT02576717) or complete the study with a safety follow-up visit 28 days after their last dose of study treatment.

ELIGIBILITY:
Inclusion Criteria:

* Multiple sclerosis as diagnosed by the revised 2010 McDonald criteria
* Expanded Disability Status Scale (EDSS) score between 0 and 5.0 at baseline

Exclusion Criteria:

* Primary progressive multiple sclerosis

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1320 (Actual)
Dates: Start 2013-12-03 (Actual); Primary Completion 2017-03-27 (Actual); Study Completion 2017-04-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (299):
- United States (35):
  - Receptos Study Site 115, Phoenix, Arizona
  - Xenoscience, Phoenix, Arizona
  - Receptos Study Site 118, Phoenix, Arizona
  - Saint Josephs Hosptial and Medical Center, Phoenix, Arizona
  - Territory Neurology and Research Institute, Tucson, Arizona
  - Receptos Study Site 119, Tucson, Arizona
  - Alta Bates Summit Medical Center, Berkeley, California
  - Receptos Study Site 110, Berkeley, California
  - Receptos Study Site 122, Long Beach, California
  - Receptos Study Site 112, Sacramento, California
  - University of California Davis Medical Center, Sacramento, California
  - Multiple Sclerosis Center at UCSF, San Francisco, California
  - Receptos Study Site 120, San Francisco, California
  - Denver Neurological Research LLC, Denver, Colorado
  - Receptos Study Site 127, Denver, Colorado
  - Neurology Associates PA, Maitland, Florida
  - Receptos Study Site 114, Maitland, Florida
  - Receptos Study Site 124, Pompano Beach, Florida
  - Neurostudies Inc, Port Charlotte, Florida
  - Receptos Study Site 123, Port Charlotte, Florida
  - Infinity Clinical Research LLC, Sunrise, Florida
  - West Georgia Sleep Disorder Center and Neurology Associates, Douglasville, Georgia
  - Consultants In Neurology, Northbrook, Illinois
  - Receptos Study Site 113, Northbrook, Illinois
  - Receptos Study Site 121, St Louis, Missouri
  - Washington University, St Louis, Missouri
  - Receptos Study Site 101, Charlotte, North Carolina
  - The Neurological Institute PA, Charlotte, North Carolina
  - Neurology and Neuroscience Associates Inc., Akron, Ohio
  - Receptos Study Site 107, Akron, Ohio
  - Receptos Study Site 104, Cleveland, Ohio
  - Receptos Study Site 109, Philadelphia, Pennsylvania
  - Receptos Study Site 102, Seattle, Washington
  - The Polyclinic, Seattle, Washington
  - Receptos Study Site 125, Tacoma, Washington
- Belarus (13):
  - Grodno Clinical Regional Hospital, Grodno
  - Receptos Study Site 907, Grodno
  - Gomel Regional Clinical Hospital, Homyel
  - Receptos Study Site 904, Homyel
  - Minsk Municipal Clinical Hospital 5, Minsk
  - Receptos Study Site 902, Minsk
  - Receptos Study Site 901, Minsk
  - Republican Scientific and Practical Centre of Neurology and Neurosurgery, Minsk
  - Minsk City Clinical Hospital 9, Minsk
  - Receptos Study Site 903, Minsk
  - Receptos Study Site 905, Vitebsk
  - Vitebsk Regional Diagnostic Centre, Vitebsk
  - Receptos Study Site 906, Vitebsk
- Belgium (8):
  - AZ Sint-Jan AV Brugge, Bruges
  - Receptos Study Site 256, Bruges
  - Cliniques Universitaires St Luc, Brussels
  - Receptos Study Site 255, Brussels
  - Centre Hospitalier Chretien Clinique Saint Joseph, Montegnée
  - Receptos Study Site 252, Montegnée
  - Clinique Saint Pierre, Ottignies
  - Receptos Study Site 254, Ottignies
- Bosnia and Herzegovina (2):
  - Clinical Center University of Sarajevo, Sarajevo
  - Receptos Study Site 911, Sarajevo
- Bulgaria (12):
  - Multiprofile Hospital for Active Treatment of Neurology and Psychiatry Sv Naum EAD, Sofia
  - Receptos Study Site 453, Sofia
  - Receptos Study Site 454, Sofia
  - Receptos Study Site 452, Sofia
  - Multiprofile Hospital for Active Treatment Tokuda Hospital Sofia, Sofia
  - Receptos Study Site 456, Sofia
  - Receptos Study Site 457, Sofia
  - University Multiprofile Hospital for Active Treatment Aleksandrovska EAD, Sofia
  - University Multiprofile Hospital for Active Treatment Sv Ivan Rilski EAD, Sofia
  - Receptos Study Site 451, Sofia
  - University Multiprofile Hospital for Active Treatment Tsaritsa Yoanna ISUL EAD, Sofia
  - Receptos Study Site 455, Sofia
- Canada (2):
  - University of Alberta MS Clinic, Edmonton, Alberta
  - Receptos Study Site 154, Edmonton, Alberta
- Croatia (8):
  - Clinical Hospital Center Osijek, Osijek
  - Receptos Study Site 923, Osijek
  - Receptos Study Site 921, Zagreb
  - Receptos Study Site 922, Zagreb
  - Receptos Study Site 924, Zagreb
  - Clinical Hospital Center "Sestre milosrdnice", Clinic of Internal Diseases, Zagreb
  - Clinical Hospital Centre Zagreb, Zagreb
  - Clinical Hospital Sveti duh, Zagreb
- Georgia (6):
  - Receptos Study Site 301, Tbilisi
  - LTD MediClubGeorgia, Tbilisi
  - Receptos Study Site 302, Tbilisi
  - Khechinashvili University Hospital, Tbilisi
  - Receptos Study Site 303, Tbilisi
  - Sarajishvili Institute of Neurology, Tbilisi
- Greece (11):
  - Evaggelismos General Hospital, Athens
  - Receptos Study Site 552, Athens
  - Receptos Study Site 554, Athens
  - Navy Hospital of Athens, Athens
  - Receptos Study Site 553, Athens
  - 401 Military Hospital of Athens, Athens
  - Receptos Study Site 551, Athens
  - AHEPA University General Hospital of Thessaloniki, Thessaloniki
  - Receptos Study Site 557, Thessaloniki
  - Georgios Papanikolaou General Hospital of Thessaloniki, Thessaloniki
  - Receptos Study Site 555, Thessaloniki
- Hungary (11):
  - Receptos Study Site 352, Budapest
  - Uzsoki Utcai Korhaz, Budapest
  - Jahn Ferenc DelPesti Korhaz es Rendelointezet, Budapest
  - Receptos Study Site 356, Budapest
  - Receptos Study Site 354, Esztergom
  - Vaszary Kolos Korhaz, Esztergom
  - Pest Megyei Flor Ferenc Korhaz, Kistarcsa
  - Receptos Study Site 358, Kistarcsa
  - Receptos Study Site 351, Nyíregyháza
  - SzabolcsSzatmarBereg Megyei Korhazak es Egyetemi Oktatokorhaz, Nyíregyháza
  - Receptos Study Site 355, Székesfehérvár
- Italy (15):
  - Azienda Ospedaliero Universitaria Policlinico Vittorio Emanuele, Catania
  - Receptos Study Site 654, Catania
  - Fondazione Istituto San Raffaele G Giglio di Cefalu, Cefalù
  - Receptos Study Site 653, Cefalù
  - Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico, Milan
  - Receptos Study Site 655, Milan
  - Receptos Study Site 652, Milan
  - Presidio Ospedaliero di Montichiari, Montichiari
  - Receptos Study Site 659, Montichiari
  - Receptos Study Site 656, Napoli
  - Receptos Study Site 658, Pavia
  - Fondazione PTV Policlinico Tor Vergata, Roma
  - Receptos Study Site 651, Roma
  - Azienda Ospedaliera Universitaria Senese, Siena
  - Receptos Study Site 657, Siena
- Moldova (5):
  - IMSP Institutul de Medicina Urgenta, Chisinau
  - Receptos Study Site 932, Chisinau
  - Institutul de Neurologie si Neurochirurgie, Chisinau
  - Receptos Study Site 931, Chisinau
  - Receptos Study Site 933, Chisinau
- Poland (52):
  - Receptos Study Site 401, Bialystok
  - Receptos Study Site 423, Bydgoszcz
  - Specjalistyczna Praktyka Lekarska Lek Med Robert Bonek, Bydgoszcz
  - Powiatowy Zespol Zakladow Opieki Zdrowotnej Szpital w Czeladzi, Czeladź
  - Receptos Study Site 406, Czeladź
  - Receptos Study Site 405, Gdansk
  - Receptos Study Site 425, Gdansk
  - Copernicus PL Sp. z. o.o., Gdansk
  - NEUROMEDIC Janusz Zbrojkiewicz, Katowice
  - MA LEK AM Maciejowscy SC Centrum Terapii SM, Katowice
  - Receptos Study Site 427, Katowice
  - NovoMed Zielinski i Wspolnicy Spolka Jawna, Katowice
  - Receptos Study Site 426, Katowice
  - NEUROCARE Site Management Organization Gabriela KlodowskaDuda, Katowice
  - Receptos Study Site 407, Katowice
  - Receptos Study Site 417, Katowice
  - Receptos Study Site 424, Kielce
  - RESMEDICA Spolka z o.o., Kielce
  - Centrum Kompleksowej Rehabilitacji Sp.z.o.o. Szpital Wielospecjalistyczny, Konstancin-Jeziorna
  - Receptos Study Site 404, Konstancin-Jeziorna
  - Krakowska Akademia Neurologii Sp. z. o.o., Krakow
  - Receptos Study Site 414, Krakow
  - Centrum Neurologii Krzysztof Selmaj, Lodz
  - Receptos Study Site 411, Lodz
  - Prof. dr med. Zbigniew Stelmasiak Specjalistyczny Gabinet Neurologiczny, Lublin
  - Receptos Study Site 412, Lublin
  - Receptos Study Site 420, Lublin
  - Wojewodzki Szpital Specjalistyczny im Stefana Kardynala Wyszynskiego, Lublin
  - Receptos Study Site 402, Olsztyn
  - Receptos Study Site 415, Olsztyn
  - Wojewodzki Szpital Specjalistyczny, Olsztyn
  - Neurologiczny NZOZ Centrum Leczenia SM Osrodek Badan Klinicznych Dr n med Hanka Hertmanowska, Plewiska
  - Receptos Study Site 421, Plewiska
  - Niepubliczny Zaklad Opieki Zdrowotnej KENDRON, Podlaskie
  - Indywidualna Specjalistyczna Praktyka Lekarska dr nmed Monika Lyczak, Pomorskie
  - Receptos Study Site 408, Poznan
  - Szpital Kliniczny im HSwiecickiego Uniwersytetu Medycznego im Karola Marcinkowskiego w Poznaniu, Poznan
  - Niepubliczny Zaklad Opieki Zdrowotnej NEUROKARD Ilkowski i Partnerzy Spolka Partnerska Lekarzy, Poznan
  - Receptos Study Site 418, Poznan
  - EUROMEDIS Sp. z.o.o., Szczecin
  - Receptos Study Site 419, Szczecin
  - Indywidualna Specjalistyczna Praktyka Lekarska Zbigniew Cebulski, Warminsko-mazurskie
  - Receptos Study Site 410, Warsaw
  - Szpital Czerniakowski Samodzielny Publiczny Zaklad Opieki Zdrowotnej, Warsaw
  - Centrum Medyczne NeuroProtect, Warsaw
  - Receptos Study Site 428, Warsaw
  - Centralny Szpital Kliniczny MSW w Warszawie, Warsaw
  - Receptos Study Site 422, Warsaw
  - Instytut Psychiatrii i Neurologii, Warsaw
  - Receptos Study Site 403, Warsaw
  - Receptos Study Site 413, Warsaw
  - Wojskowy Instytut Medyczny, Warsaw
- Romania (10):
  - Clinical Hospital of Psychiatry and Neurology Brasov, Brasov
  - Receptos Study Site 503, Brasov
  - Health Club Medical Center S.R.L., Campulung Muscel
  - Receptos Study Site 502, Campulung Muscel
  - Receptos Study Site 501, Cluj-Napoca
  - Rehabilitation Clinical Hospital, Cluj-Napoca
  - Receptos Study Site 505, Sibiu
  - Sibiu Emergency County Clinical Hospital, Sibiu
  - Receptos Study Site 506, Timișoara
  - Timisoara Emergency County Clinical Hospital, Timișoara
- Russia (28):
  - Chelyabinsk City Clinical Hospital 3, Chelyabinsk
  - Receptos Study Site 701, Chelyabinsk
  - Receptos Study Site 704, Kazan'
  - Republican Clinical Hospital for Rehabilitation Treatment, Kazan'
  - Receptos Study Site 713, Kazan'
  - Research Medical Complex Vashe Zdorovie, Kazan'
  - Central Clinical Hospital 2 na NA Semashko OAO RZhD, Moscow
  - Receptos Study Site 712, Moscow
  - City Clinical Hospital 1 na NIPirogov, Moscow
  - Receptos Study Site 709, Moscow
  - City neurology center Sibneuromed LLC, Novosibirsk
  - Receptos Study Site 703, Novosibirsk
  - Perm State Medical Academy, Perm
  - Receptos Study Site 710, Perm
  - Receptos Study Site 708, Saint Petersburg
  - Russian Medical Military Academy na SMKirov, Saint Petersburg
  - Receptos Study Site 716, Samara
  - Samara Regional Clinical Hospital named after MI Kalinin, Samara
  - City Clinical Hospital 4, Saransk
  - Receptos Study Site 715, Saransk
  - Receptos Study Site 714, Saratov
  - Saratov State Medical University, Saratov
  - Receptos Study Site 707, Smolensk
  - Smolensk State Medical Academy, Smolensk
  - Receptos Study Site 717, Tyumen
  - Neftyanik Medical and Sanitary Unit, Tyumen
  - Receptos Study Site 711, Yaroslavl
  - Yaroslavl Clinical Hospital 8, Yaroslavl
- Serbia (10):
  - Clinical Center of Serbia, Belgrade
  - Clinical Hospital Centar Zvezdara, Belgrade
  - Military Medical Academy, Belgrade
  - Receptos Study Site 602, Belgrade
  - Receptos Study Site 603, Belgrade
  - Receptos Study Site 604, Belgrade
  - Clinical Hospital Centre Zemun, Belgrade
  - Receptos Study Site 601, Belgrade
  - Clinical Center Kragujevac, Kragujevac
  - Receptos Study Site 605, Kragujevac
- Slovakia (4):
  - University Hospital Bratislava - Hospital ak. L. Derera, II Neurology Clinic, Bratislava
  - Receptos Study Site 946, Bratislava
  - Receptos Study Site 942, Lučenec
  - Receptos Study Site 945, Trnava
- South Africa (3):
  - Receptos Study Site 956, KwaZulu-Natal
  - Neurology Practice, Pretoria
  - Receptos Study Site 953, Pretoria
- Spain (21):
  - Receptos Study Site 755, Seville, Andalusia
  - Receptos Study Site 761, Bilbao, Basque Country
  - Receptos Study Site 759, Donostia / San Sebastian, Basque Country
  - Receptos Study Site 763, Santa Cruz de Tenerife, Canary Islands
  - Receptos Study Site 756, Barcelona, Catalonia
  - Receptos Study Site 760, Girona, Catalonia
  - Receptos Study Site 762, Alicante, Valencia
  - Receptos Study Site 752, Valencia, Valencia
  - Hospital General Universitario de Alicante, Alicante
  - Hospital del Mar, Barcelona
  - Receptos Study Site 758, Barcelona
  - Hospital Universitario Vall D hebron, Barcelona
  - Organizacion Sanitaria Integrada Bilbao Basurto, Bilbao
  - Hospital Universitari de Girona Dr Josep Trueta, Girona
  - Hospital Universitario de la Princesa, Madrid
  - Receptos Study Site 757, Madrid
  - Receptos Study Site 751, Madrid
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda
  - Receptos Study Site 754, Majadahonda (Madrid)
  - Hospital Universitario Vírgen Macarena, Seville
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia
- Ukraine (32):
  - Municipal Medical & Preventive Institution Chernigiv Regional Clinical Hospital, Chernihiv
  - Receptos Study Site 805, Chernihiv
  - Municipal Institution Chernivtsi Regional Psychiatric Hospital, Chernivtsi
  - Receptos Study Site 813, Chernivtsi
  - Municipal Institution Dnipropetrovsk Regional Clinical Hospital na I.I. Mechnykov, Dnipropetrovsk
  - Receptos Study Site 802, Dnipropetrovsk
  - State Institution Dnipropetrovsk Medical Academy of the Ministry of Health of Ukraine, Dnipropetrovsk
  - Receptos Study Site 815, Dnipropetrovsk
  - Receptos Study Site 801, Ivano-Frankivsk
  - Regional Clinical Hospital, Ivano-Frankivsk
  - Receptos Study Site 814, Kharkiv
  - State Treatment and Prevention Institution Central Clinical Hospital of Ukrzaliznytsya, Kharkiv
  - Municipal Institution Kherson City Clinical Hospital, Kherson
  - Receptos Study Site 811, Kherson
  - Receptos Study Site 818, Kyiv
  - Municipal Institution of Kyiv Regional Council Kyiv Regional Clinical Hospital, Kyiv
  - Receptos Study Site 803, Kyiv
  - Kyiv City Clinical Hospital 4, Kyiv
  - Municipal Institution Lutsk City Clinical Hospital, Lutsk
  - Receptos Study Site 816, Lutsk
  - Receptos Study Site 817, Lutsk
  - Volyn Regional Clinical Hospital, Lutsk
  - Lviv Regional Clinical Hospital, Lviv
  - Receptos Study Site 812, Lviv
  - Center for Reconstructive and Rehabilitation Medicine University Clinic of ONMedU, Odesa
  - Receptos Study Site 810, Odesa
  - Municipal Institution Odesa Regional Clinical Hospital, Odesa
  - Receptos Study Site 804, Odesa
  - Municipal Institution Vinnytsya Regional Psychoneurological Hospital na OI Yushchenko, Vinnytsia
  - Receptos Study Site 809, Vinnytsia
  - Municipal Institution City Clinical Hospital 6, Zaporizhzhya
  - Receptos Study Site 806, Zaporizhzhya
- United Kingdom (11):
  - Receptos Study Site 965, Brighton
  - Royal Sussex County Hospital, Brighton East Sussex
  - Raigmore Hospital, Inverness
  - Receptos Study Site 963, Inverness
  - Kings College Hospital, London
  - Receptos Study Site 961, London
  - National Hospital for Neurology and Neurosurgery, London
  - Receptos Study Site 967, London
  - Receptos Study Site 966, Romford
  - Receptos Study Site 964, Sheffield
  - Royal Hallamshire Hospital Sheffield Teaching Hospitals NHS Trust, Sheffield

REFERENCES:
- [Result] Cree B, et al. The RADIANCE and SUNBEAM phase 3 studies of ozanimod in relapsing multiple sclerosis: study design and baseline characteristics. Presented at the 69th Annual American Academy of Neurology Meeting, April 22-28, 2017, Boston, MA. Abstract No. P6-344
- [Result] Cohen JA, Comi G, Selmaj KW, Bar-Or A, Arnold DL, Steinman L, Hartung HP, Montalban X, Kubala Havrdova E, Cree BAC, Sheffield JK, Minton N, Raghupathi K, Huang V, Kappos L; RADIANCE Trial Investigators. Safety and efficacy of ozanimod versus interferon beta-1a in relapsing multiple sclerosis (RADIANCE): a multicentre, randomised, 24-month, phase 3 trial. Lancet Neurol. 2019 Nov;18(11):1021-1033. doi: 10.1016/S1474-4422(19)30238-8. Epub 2019 Sep 3. PMID 31492652
- [Derived] Harris S, Comi G, Cree BAC, Arnold DL, Steinman L, Sheffield JK, Maddux R, Southworth H, Kappos L, Cohen JA. Glial Fibrillary Acidic Protein as a Marker of Disease in Relapsing Multiple Sclerosis: Post Hoc Analysis of Phase 3 Ozanimod Trials. Eur J Neurol. 2025 Jun;32(6):e70222. doi: 10.1111/ene.70222. PMID 40462564

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 147 academic medical centers and clinical practices in 21 countries in North America, Europe, and South Africa. Between December 2013 and March 2015, 1695 participants were screened, of which 375 did not meet inclusion criteria. One thousand, three hundred and twenty participants with relapsing multiple sclerosis (MS) were enrolled and randomly assigned to a treatment group.
Pre-assignment Details: Participants were randomized in a 1:1:1 ratio to one of three treatment groups. Randomization was stratified by Baseline Expanded Disability Status Scale (EDSS) score (≤ 3.5, > 3.5) and by country.
  Participants who completed the 24-month study were eligible to enroll in a long-term, open-label extension study (RPC01-3001; NCT02576717).
Groups:
- Interferon Beta-1a (IFN β-1a): Participants received interferon beta-1a (IFN β-1a) 30 µg intramuscular (IM) injection weekly and matching placebo capsules (identical in physical appearance to ozanimod) orally daily for 24 months.
- Ozanimod 0.5 mg: Participants received ozanimod 0.5 mg oral capsules daily and an intramuscular placebo injection (identical in appearance to Interferon) weekly for 24 months.
- Ozanimod 1 mg: Participants received ozanimod 1 mg oral capsules daily and an intramuscular placebo injection (identical in appearance to interferon) weekly for 24 months.
Period: Overall Study
Arm/Group | Interferon Beta-1a (IFN β-1a) | Ozanimod 0.5 mg | Ozanimod 1 mg
Started | 443 | 443 | 434
Received Treatment | 441 (One participant received ozanimod 0.5 mg in error) | 439 (One participant received ozanimod 1.0 mg in error) | 433
Completed (Completed study drug) | 376 | 374 | 388
Not Completed | 67 | 69 | 46
Not completed — Adverse Event | 18 | 13 | 13
Not completed — Lack of Efficacy | 4 | 5 | 1
Not completed — Protocol Violation | 3 | 1 | 1
Not completed — Lost to Follow-up | 1 | 4 | 0
Not completed — Death | 0 | 1 | 0
Not completed — Withdrawal by Subject | 30 | 31 | 19
Not completed — Physician Decision | 7 | 6 | 5
Not completed — Miscellaneous | 2 | 4 | 6
Not completed — Did Not Receive Study Drug | 2 | 4 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all randomized participants who received at least 1 dose of study drug; participants were analyzed according to the treatment they were randomized to receive and not according to what they actually received, if different.
Groups:
- Interferon Beta-1a (IFN β-1a): Participants received IFN β-1a 30 µg intramuscular (IM) injection weekly and matching placebo capsules (identical in physical appearance to ozanimod) orally daily for 24 months.
- Total: Total of all reporting groups
Arm/Group | Interferon Beta-1a (IFN β-1a) | Ozanimod 0.5 mg | Ozanimod 1 mg | Total
Number analyzed (Participants) | 441 | 439 | 433 | 1313
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.1 (9.07) | 35.4 (8.82) | 36.0 (8.89) | 35.5 (8.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 304 | 287 | 291 | 882
  Male | 137 | 152 | 142 | 431
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 6 | 10 | 21
  Not Hispanic or Latino | 436 | 433 | 423 | 1292
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 432 | 431 | 428 | 1291
  Black | 7 | 6 | 5 | 18
  Asian | 1 | 0 | 0 | 1
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Other | 1 | 2 | 0 | 3
Region [Count of Participants; unit: Participants]
  North America | 16 | 16 | 16 | 48
  Western Europe | 40 | 40 | 36 | 116
  Eastern Europe | 379 | 378 | 374 | 1131
  Southern Africa | 6 | 5 | 7 | 18
Country of Enrollment [Count of Participants; unit: Participants]
  Belarus | 40 | 38 | 37 | 115
  Belgium | 4 | 4 | 4 | 12
  Bosnia And Herzegovina | 3 | 3 | 2 | 8
  Bulgaria | 11 | 12 | 11 | 34
  Canada | 1 | 1 | 0 | 2
  Croatia | 16 | 15 | 14 | 45
  Georgia | 12 | 11 | 13 | 36
  Greece | 3 | 4 | 2 | 9
  Hungary | 7 | 9 | 6 | 22
  Italy | 8 | 9 | 7 | 24
  Poland | 125 | 124 | 124 | 373
  Republic of Moldova | 2 | 4 | 3 | 9
  Romania | 9 | 9 | 10 | 28
  Russian Federation | 41 | 40 | 40 | 121
  Serbia | 34 | 34 | 34 | 102
  Slovakia | 2 | 1 | 2 | 5
  South Africa | 6 | 5 | 7 | 18
  Spain | 19 | 17 | 19 | 55
  Ukraine | 77 | 78 | 78 | 233
  United Kingdom | 6 | 6 | 4 | 16
  United States | 15 | 15 | 16 | 46
Type of Multiple Sclerosis [Count of Participants; unit: Participants]
  Relapsing-remitting multiple sclerosis | 432 | 432 | 425 | 1289
  Progressive-relapsing multiple sclerosis | 8 | 7 | 8 | 23
  Secondary progressive multiple sclerosis | 1 | 0 | 0 | 1
Age at MS Symptom Onset [Mean (Standard Deviation); unit: years] | 28.9 (8.60) | 29.3 (8.41) | 29.2 (8.67) | 29.1 (8.56)
Age at MS Diagnosis [Mean (Standard Deviation); unit: years] | 31.6 (8.82) | 32.0 (8.59) | 32.1 (8.95) | 31.9 (8.78)
Time Since MS Symptom Onset [Mean (Standard Deviation); unit: years] | 6.36 (6.065) | 6.23 (5.547) | 6.92 (6.201) | 6.50 (5.947)
Expanded Disability Status Scale (EDSS) Score [Mean (Standard Deviation); unit: units on a scale] — The EDSS is a scale for quantifying disability in MS. Eight functional systems (visual, brain stem, pyramidal, cerebellar, sensory, bowel & bladder, cerebral, and other functions) are scored on a scale from 0 (no disability) to 5 or 6 (more severe disability). Ambulation is also scored. Based on scores in the 8 functional systems plus gait, an overall score ranging from 0 (normal) to 10 (death due to MS) in 0.5 unit increments is assigned. Participants with EDSS scores of 0.0 to 4.5 are fully ambulatory; patients with EDSS scores of 5.0 to 9.5 have impaired ambulation.
  units on a scale | 2.49 (1.158) | 2.48 (1.166) | 2.55 (1.145) | 2.51 (1.156)
EDSS Category [Count of Participants; unit: Participants] — The EDSS is a scale for quantifying disability in MS. Eight functional systems (visual, brain stem, pyramidal, cerebellar, sensory, bowel & bladder, cerebral, and other functions) are scored on a scale of 0 (no disability) to 5 or 6 (more severe disability). Ambulation is also scored. Based on scores in these 8 functional systems and gait, an overall score ranging from 0 (normal) to 10 (death due to MS) in 0.5 unit increments is assigned. Participants with EDSS scores of 0.0 to 4.5 are fully ambulatory; patients with EDSS scores of 5.0 to 9.5 have impaired ambulation.
  Participants
    EDSS ≤ 3.5 | 375 | 374 | 371 | 1120
    EDSS > 3.5 | 66 | 65 | 62 | 193
Number of Gadolinium-enhancing (GdE) Lesions [Mean (Standard Deviation); unit: lesions] — A lesion appearing on magnetic resonance imagery (MRI), following injection of the chemical compound gadolinium, that reveals a breakdown in the blood-brain barrier. This breakdown of the blood-brain barrier indicates either a newly active lesion or the re-activation of an old one. Population: Participants with available MRI data
  lesions
    number analyzed (Participants) | 440 | 439 | 433 | 1312
    (all) | 1.8 (3.54) | 1.8 (3.62) | 1.6 (3.78) | 1.7 (3.65)
Number of T2 Lesions [Mean (Standard Deviation); unit: lesions] — A T2-weighted MRI scan shows the number of old and new lesions in a specific part of the brain or spinal cord. Population: Participants with available MRI data
  lesions
    number analyzed (Participants) | 440 | 439 | 432 | 1311
    (all) | 48.7 (32.62) | 48.7 (36.27) | 47.9 (32.37) | 48.4 (33.78)
Normalized Brain Volume [Mean (Standard Deviation); unit: cm³] — Measured using MRI Population: Participants with available data
  cm³
    number analyzed (Participants) | 439 | 437 | 432 | 1308
    (all) | 1449.581 (77.156) | 1452.852 (71.978) | 1441.949 (79.228) | 1448.153 (76.250)

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Annualized Relapse Rate (ARR) at the End of Month 24
Description: A relapse was defined as new or worsening neurological symptoms attributable to MS and preceded by a relatively stable or improving neurological state for at least 30 days. Symptoms must have persisted for > 24 hours and not be attributable to confounding clinical factors. Relapses were confirmed when accompanied by objective neurological worsening based on examination by the blinded evaluator, consistent with an increase of ≥ 0.5 on the overall EDSS score relative to the most recent EDSS assessment, or 2 points on one of the functional system scale scores, or 1 point on ≥ two functional system scale scores.
  Relapse rate was calculated as the total number of confirmed relapses divided by the total number of days in the study * 365.25.
  ARR was based on a Poisson regression model, adjusted for region (Eastern Europe vs Rest of the World), age, and the Baseline number of gadolinium-enhancing lesions, and included the natural log transformation of time on study as an offset term.
Time Frame: At the end of month 24
Population: The ITT population included all randomized participants who received at least 1 dose of study drug; participants were analyzed according to the treatment they were randomized to receive and not according to what they actually received, if different.
Measure: Number (95% Confidence Interval); unit: relapses/year
Groups:
- Interferon Beta-1a: Participants received IFN β-1a 30 µg intramuscular injection weekly and matching placebo capsules (identical in physical appearance to ozanimod) orally daily for 24 months.
Arm/Group | Interferon Beta-1a | Ozanimod 0.5 mg | Ozanimod 1 mg
Number analyzed (Participants) | 441 | 439 | 433
relapses/year | 0.276 [0.234 to 0.324] | 0.218 [0.183 to 0.259] | 0.172 [0.142 to 0.208]
Statistical Analysis 1: Comparison: Interferon Beta-1a vs Ozanimod 1 mg; Test type: Superiority; p < 0.0001, Poisson regression model — To account for multiple comparisons, each of the 2 treatment comparisons was tested at the alpha = 0.025 level; Adjusted for region, age, and Baseline number of GdE lesions, and Included the natural log transformation of time on study as an offset term; Rate Ratio = 0.623, 95% CI 2-sided [0.506 to 0.768] — Rate Ratio = Ozanimod / IFN β-1a
Statistical Analysis 2: Comparison: Interferon Beta-1a vs Ozanimod 0.5 mg; Test type: Superiority; p = 0.0167, Poisson Regression Model — To account for multiple comparisons, each of the 2 treatment comparisons was tested at the alpha = 0.025 level; [statistical method as in outcome 1, analysis 1]; Rate Ratio = 0.791, 95% CI 2-sided [0.652 to 0.958] — Rate Ratio = Ozanimod / IFN β-1a

2. Secondary Outcome: Adjusted Mean Number of New or Enlarging Hyperintense T2-Weighted Brain Magnetic Resonance Imaging (MRI) Lesions Per Scan Over 24 Months
Description: The adjusted mean number of new or enlarging hyperintense T2-weighted brain MRI lesions per scan was based on the cumulative number of new or enlarging T2 lesions since Baseline over 24 months. MRI images were assessed and scored by an independent MRI analysis center with no knowledge of treatment assignment or outcomes.
  The adjusted mean per scan over 24 months was based based on a negative binomial regression model using observed data, adjusted for region (Eastern Europe vs. Rest of the World), age at Baseline, and Baseline number of GdE lesions. The natural log transformation of the number of available MRI scans over 24 months is used as an offset term.
Time Frame: 24 month treatment period; MRI scans were performed at Months 12 and 24
Population: ITT Population included all randomized participants who received at least 1 dose of study drug. Includes participants with non-missing MRI results.
Measure: Least Squares Mean (95% Confidence Interval); unit: lesions/scan
Arm/Group | Interferon Beta-1a | Ozanimod 0.5 mg | Ozanimod 1 mg
Number analyzed (Participants) | 336 | 329 | 327
lesions/scan | 3.183 [2.640 to 3.838] | 2.092 [1.741 to 2.514] | 1.835 [1.523 to 2.211]
Statistical Analysis 1: Comparison: Interferon Beta-1a vs Ozanimod 1 mg; Test type: Superiority; p < 0.0001, Negative Binomial Regression Model — To control for type 1 error, the key secondary endpoints were tested in order in a sequential, closed hierarchical testing procedure. Each comparison was tested at the alpha = 0.05 level; Adjusted for region, age, and Baseline GdE lesions, and included the natural log transformation of available number of MRI scans as an offset term; Rate Ratio = 0.576, 95% CI 2-sided [0.465 to 0.714] — Rate Ratio = Ozanimod / IFN β-1a
Statistical Analysis 2: Comparison: Interferon Beta-1a vs Ozanimod 0.5 mg; Test type: Superiority; p = 0.0001, Negative binomial regression model — [p-value comment as in outcome 2, analysis 1]; Adjusted for region, age, and Baseline GdE lesions and included the natural log transformation of available number of MRI scans as an offset term; Rate Ratio = 0.657, 95% CI 2-sided [0.531 to 0.813] — Rate Ratio = Ozanimod / IFN β-1a

3. Secondary Outcome: Adjusted Mean Number of Gadolinium Enhancing Brain Lesions at Month 24
Description: MRI images were assessed and scored by an independent MRI analysis center with no knowledge of treatment assignment or outcomes.
  The number of gadolinium-enhancing (GdE) lesions at 24 months was analyzed based on observed data using a negative binomial regression model adjusted for region (Eastern Europe vs Rest of World), Baseline age, and Baseline number of GdE lesions, with natural log transformation of number of available MRI scans over 24 months as an offset term (1 scan for per participant).
Time Frame: Month 24
Population: The ITT population consisted of all randomized participants who received at least 1 dose of study medication. Includes participants with non-missing GdE MRI results at Month 24.
Measure: Least Squares Mean (95% Confidence Interval); unit: lesions
Arm/Group | Interferon Beta-1a | Ozanimod 0.5 mg | Ozanimod 1 mg
Number analyzed (Participants) | 336 | 329 | 327
lesions | 0.373 [0.256 to 0.543] | 0.197 [0.131 to 0.296] | 0.176 [0.116 to 0.266]
Statistical Analysis 1: Comparison: Interferon Beta-1a vs Ozanimod 1 mg; Test type: Superiority; p = 0.0006, Negative Binomial Regression Model — [p-value comment as in outcome 2, analysis 1]; Adjusted for region, age, and Baseline GdE lesions with the natural log transformation of available MRI scans at Month 24 as an offset term; Rate Ratio = 0.471, 95% CI 2-sided [0.306 to 0.725] — Rate ratio = Ozanimod / IFN β-1a
Statistical Analysis 2: Comparison: Interferon Beta-1a vs Ozanimod 0.5 mg; Test type: Superiority; p = 0.0030, Negative binomial regression model, — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 3, analysis 1]; Rate Ratio = 0.528, 95% CI 2-sided [0.346 to 0.805] — Rate ratio = Ozanimod / IFN β-1a

4. Secondary Outcome: Time to Onset of Disability Progression Confirmed After 3 Months
Description: EDSS is used to quantify disability and disability progression over time in MS. Based on a neurological examination, 8 functional systems (visual, brain stem, pyramidal, cerebellar, sensory, bowel & bladder, cerebral, and other functions) are scored from 0 (no disability) to 5 or 6 (more severe disability). Ambulation is assessed based on distance the patient is able to walk, whether assistance is required or restrictions are present.
  The EDSS score ranges from 0 (normal) to 10 (death due to MS) in 0.5 unit increments.
  Disability progression is defined by a sustained worsening in EDSS score of 1.0 point or more confirmed after 3 months. Time to onset of disability progression was calculated from the date of first dose to the date of the first visit at which the 1.0 point increase in EDSS was met using Kaplan-Meier methods. Participants without a sustained disease progression event were censored on the date of their last assessment or last dose of study drug, whichever was later.
Time Frame: From first dose to the end of the 24-month treatment period
Population: The ITT population consisted of all randomized participants who received at least 1 dose of study medication.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Interferon Beta-1a | Ozanimod 0.5 mg | Ozanimod 1 mg
Number analyzed (Participants) | 441 | 439 | 433
days | NA [NA to NA] — Not estimable as there were insufficient disability events | NA [NA to NA] — Not estimable as there were insufficient disability events | NA [NA to NA] — Not estimable as there were insufficient disability events
Statistical Analysis 1: Comparison: Interferon Beta-1a vs Ozanimod 1 mg; Test type: Superiority; p = 0.8224, Cox proportional hazards model — [p-value comment as in outcome 2, analysis 1]; Adjusted for region (Eastern Europe vs Rest of World) age at Baseline, and Baseline EDSS score; Hazard Ratio (HR) = 1.045, 95% CI 2-sided [0.711 to 1.537] — Hazard ratio (Ozanimod / IFN β-1a) based on Cox proportional hazard model with factors for treatment group, adjusted for region, age at Baseline, and Baseline EDSS score
Statistical Analysis 2: Comparison: Interferon Beta-1a vs Ozanimod 0.5 mg; Test type: Superiority; p = 0.2849, Cox proportional hazards model — [p-value comment as in outcome 2, analysis 1]; Adjusted for region (Eastern Europe vs Rest of World), age at Baseline, and Baseline EDSS score; Hazard Ratio (HR) = 0.798, 95% CI 2-sided [0.528 to 1.206] — [estimate comment as in outcome 4, analysis 1]

5. Secondary Outcome: Time to Onset of Disability Progression Confirmed After 6 Months
Description: as for outcome 4
Time Frame: From first dose to the end of the 24-month treatment period
Population: The ITT population consisted of all randomized participants who received at least 1 dose of study medication.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Interferon Beta-1a | Ozanimod 0.5 mg | Ozanimod 1 mg
Number analyzed (Participants) | 441 | 439 | 433
days | NA [NA to NA] — Not estimable as there were insufficient disability events | NA [NA to NA] — Not estimable as there were insufficient disability events | NA [NA to NA] — Not estimable as there were insufficient disability events
Statistical Analysis 1: Comparison: Interferon Beta-1a vs Ozanimod 1 mg; Test type: Superiority; p = 0.1353, Cox proportional hazard model — [p-value comment as in outcome 2, analysis 1]; Adjusted for region (Eastern Europe vs Rest of World), age at Baseline, and Baseline EDSS score; Hazard Ratio (HR) = 1.435, 95% CI 2-sided [0.893 to 2.305] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Interferon Beta-1a vs Ozanimod 0.5 mg; Test type: Superiority; p = 0.7154, Cox proportional hazard model — [p-value comment as in outcome 2, analysis 1]; Adjusted for region (Eastern Europe vs Rest of World), age at Baseline, and Baseline EDSS score; Hazard Ratio (HR) = 1.098, 95% CI 2-sided [0.664 to 1.815] — [estimate comment as in outcome 4, analysis 1]

6. Secondary Outcome: Percentage of Participants Who Were Gadolinium Enhancing (GdE) Lesion-Free at Month 24
Description: Participants were considered lesion free at Month 24 if they did not show evidence of GdE lesions at the Month 24 MRI scan.
  MRI images were assessed and scored by an independent MRI analysis center with no knowledge of treatment assignment or outcomes.
Time Frame: Month 24
Population: ITT population included all randomized participants who received at least 1 dose of study drug; participants with missing data at Month 24 were considered non-responders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Interferon Beta-1a | Ozanimod 0.5 mg | Ozanimod 1 mg
Number analyzed (Participants) | 441 | 439 | 433
percentage of participants | 56.2 [51.6 to 60.9] | 63.3 [58.8 to 67.8] | 65.6 [61.1 to 70.1]
Statistical Analysis 1: Comparison: Interferon Beta-1a vs Ozanimod 1 mg; Test type: Superiority; p = 0.0047, Cochran-Mantel-Haenszel; Stratified by region (Eastern Europe vs Rest of the World) and Baseline EDSS category; Difference = 9.4, 95% CI 2-sided [2.9 to 15.8]
Statistical Analysis 2: Comparison: Interferon Beta-1a vs Ozanimod 0.5 mg; Test type: Superiority; p = 0.0320, Cochran-Mantel-Haenszel; Stratified by region (Eastern Europe vs Rest of the World) and Baseline EDSS category; Difference = 7.1, 95% CI 2-sided [0.6 to 13.6]

7. Secondary Outcome: Percentage of Participants Who Were New or Enlarging T2 Lesion-Free at Month 24
Description: MRI images were assessed and scored by an independent MRI analysis center with no knowledge of treatment assignment or outcomes.
Time Frame: Month 24
Population: The ITT population consisted of all randomized participants who received at least 1 dose of study medication; Participants with missing data at Month 24 were considered non-responders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Interferon Beta-1a | Ozanimod 0.5 mg | Ozanimod 1 mg
Number analyzed (Participants) | 441 | 439 | 433
percentage of participants | 18.4 [14.8 to 22.0] | 23.5 [19.5 to 27.4] | 23.8 [19.8 to 27.8]
Statistical Analysis 1: Comparison: Interferon Beta-1a vs Ozanimod 1 mg; Test type: Superiority; p = 0.0466, Cochran-Mantel-Haenszel; Based on the Cochran-Mantel-Haenszel test stratified by region (Eastern Europe vs. rest of the world) and Baseline EDSS category; Difference = 5.4, 95% CI 2-sided [0.0 to 10.8]
Statistical Analysis 2: Comparison: Interferon Beta-1a vs Ozanimod 1 mg; Test type: Superiority; p = 0.0581, Cochran-Mantel-Haenszel; [statistical method as in outcome 7, analysis 1]; Difference = 5.1, 95% CI 2-sided [-0.3 to 10.5]

8. Secondary Outcome: Percent Change From Baseline in Normalized Brain Volume to Month 24
Description: Brain volume (a measure of brain atrophy) was measured by brain MRI scans that were assessed and scored by an independent MRI analysis center with no knowledge of treatment assignment or outcomes.
Time Frame: Baseline and Month 24
Population: ITT Population; last observation carried forward was used for participants with missing data at Month 24 (only post-baseline MRI scans were carried forward)
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Interferon Beta-1a | Ozanimod 0.5 mg | Ozanimod 1 mg
Number analyzed (Participants) | 397 | 398 | 390
percent change | -0.937 (0.944) | -0.707 (0.746) | -0.707 (0.878)
Statistical Analysis 1: Comparison: Interferon Beta-1a vs Ozanimod 1 mg; Test type: Superiority; p < 0.0001, ANCOVA — Based on the analysis of covariance model, adjusted for region (Eastern Europe vs. rest of the world), Baseline EDSS category, and brain volume at Baseline; Difference in means = 0.244, 95% CI 2-sided [0.125 to 0.363] — Difference in means based on the analysis of covariance model, adjusted for region (Eastern Europe vs. rest of the world), Baseline EDSS category, and brain volume at Baseline
Statistical Analysis 2: Comparison: Interferon Beta-1a vs Ozanimod 0.5 mg; Test type: Superiority; p = 0.0002, ANCOVA — [p-value comment as in outcome 8, analysis 1]; Difference in means = 0.224, 95% CI 2-sided [0.106 to 0.342] — [estimate comment as in outcome 8, analysis 1]

9. Secondary Outcome: Change From Baseline to Month 24 in Multiple Sclerosis Functional Composite (MSFC) Score Including the Low-Contrast Letter Acuity (LCLA) Test
Description: The MSFC-LCLA is a battery including the following 4 individual scales:
  * Timed 25-Foot Walk is an ambulation measure of walking 25 feet with time taken recorded in seconds
  * 9-Hole Peg Test (9HPT) is a quantitative measure of upper extremity (arm and hand) function
  * Symbol Digit Modalities Test (SDMT) is a measure of executive cognitive function that assesses processing speed, flexibility, and calculation ability
  * Low-Contrast Letter Acuity Test (LCLA) used a standardized set of charts to assess low contrast visual acuity, charts are scored according to the number of letters that are identified correctly
  Z-scores were calculated for for each component and averaged to create an overall composite score, using the study population as the reference population. A Z-score represents the number of standard deviations a patient's test result is higher (Z > 0) or lower (Z < 0) than the average test result (Z = 0) of the reference population. A positive change indicates improvement.
Time Frame: Baseline to Month 24
Population: The ITT population with available MSFC Z-scores
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Interferon Beta-1a | Ozanimod 0.5 mg | Ozanimod 1 mg
Number analyzed (Participants) | 437 | 435 | 428
Z-score | -0.052 (0.601) | 0.036 (0.440) | -0.010 (0.622)
Statistical Analysis 1: Comparison: Interferon Beta-1a vs Ozanimod 1 mg; Test type: Superiority; p = 0.2480, ANCOVA; Based on the analysis of covariance model, adjusted for region, Baseline EDSS category, and Baseline MSFC Z-score; Difference in means = 0.043, 95% CI 2-sided [-0.030 to 0.116] — Difference in means are based on the analysis of covariance model, adjusted for region (Eastern Europe vs Rest of the World), Baseline EDSS category, and the Baseline MSFC Z-score
Statistical Analysis 2: Comparison: Interferon Beta-1a vs Ozanimod 0.5 mg; Test type: Superiority; p = 0.0123, ANCOVA; Based on the analysis of covariance model, adjusted for region, Baseline EDSS category, and Baseline MSFC Z-score; Difference in means = 0.093, 95% CI 2-sided [0.020 to 0.165] — Difference in means based on the analysis of covariance model, adjusted for region (Eastern Europe vs Rest of the World), Baseline EDSS category, and the Baseline MSFC Z-score

10. Secondary Outcome: Mean Change From Baseline in Multiple Sclerosis Quality of Life (MSQOL)-54 Physical Health Composite Summary and Mental Health Composite Summary Scores
Description: The MSQOL-54 is a multidimensional health-related QOL measure that combines both generic and MS-specific items into a single instrument. The instrument includes 12 subscales, two summary scores, and two single-item measures.
  The two summary scores - physical health and mental health - are derived from a weighted combination of scale scores.
  The physical health composite score includes Physical function, Health perceptions, Energy/fatigue, Role limitations - physical, Pain, Sexual function, Social function, and Health distress.
  The mental health composite score includes Health distress, Overall quality of life, Emotional well-being, Role limitations - emotional, and Cognitive function.
  Each composite summary score has a range from 0 to 100 where higher scores indicate better quality of life. A positive change from Baseline indicates improvement.
Time Frame: Baseline to Month 24
Population: The ITT population consisted of all randomized participants who received at least 1 dose of study medication. Missing data were imputed using a mixed-effects regression model.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Interferon Beta-1a | Ozanimod 0.5 mg | Ozanimod 1 mg
Number analyzed (Participants) | 441 | 439 | 433
units on a scale
  Physical Health Composite Summary | -1.526 (12.319) | 0.609 (12.315) | 0.209 (12.321)
  Mental Health Composite Summary | -1.831 (16.422) | -1.182 (14.379) | -1.517 (15.544)
Statistical Analysis 1: Comparison: Interferon Beta-1a vs Ozanimod 1 mg; Analysis of Physical Health Composite Summary Score; Test type: Superiority; p = 0.0988, ANCOVA; Based on the analysis of covariance model, adjusted for region, Baseline EDSS category, and Baseline summary score; Difference in means = 1.345, 95% CI 2-sided [-0.252 to 2.943] — Difference in means based on the analysis of covariance model, adjusted for region (Eastern Europe vs Rest of the World), Baseline EDSS category, and Baseline summary score
Statistical Analysis 2: Comparison: Interferon Beta-1a vs Ozanimod 0.5 mg; Analysis of Physical Health Composite Summary Score; Test type: Superiority; p = 0.0228, ANCOVA; Based on the analysis of covariance model, adjusted for region, Baseline EDSS category, and Baseline summary score; Difference in means = 1.849, 95% CI 2-sided [0.258 to 3.440] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: Interferon Beta-1a vs Ozanimod 1 mg; Analysis of Mental Health Composite Summary Score; Test type: Superiority; p = 0.6997, ANCOVA; Based on the analysis of covariance model, adjusted for region, Baseline EDSS category, and Baseline summary score; Difference in means = 0.380, 95% CI 2-sided [-1.553 to 2.313] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 4: Comparison: Interferon Beta-1a vs Ozanimod 0.5 mg; Analysis of Mental Health Composite Summary Score; Test type: Superiority; p = 0.5501, ANCOVA; Based on the analysis of covariance model, adjusted for region, Baseline EDSS category, and the Baseline summary score; Difference in means = 0.587, 95% CI 2-sided [-1.339 to 2.513] — [estimate comment as in outcome 10, analysis 1]

11. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events
Description: An adverse event (AE) is any untoward medical occurrence that does not necessarily have a causal relationship with the investigational product (IP), including an abnormal laboratory finding, symptom or disease temporally associated with the use of an IP whether or not considered related to the IP. Serious AEs were events that resulted in death, were life-threatening, required hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability or incapacity, were congenital abnormalities/birth defects, or important medical events which may have required medical intervention to prevent one of the above outcomes.
  The investigator assessed the severity of AEs as mild, moderate, or severe and the relationship of each AE to treatment as unrelated, unlikely, possible, probable, or related based on timing and other known factors such as clinical state, environment, or other therapies.
Time Frame: From the first dose of study drug up to the first dose of the open-label extension study RPC01-3001, or up to 28 days after last dose for participants who did not continue into the open-label extension study; median duration of treatment was 24 months.
Population: Safety Population included all participants who received at least 1 dose of study drug, analyzed according to the highest dose of ozanimod treatment actually received, not according to the treatment they were randomized to receive, if different.
Measure: Count of Participants; unit: Participants
Arm/Group | Interferon Beta-1a | Ozanimod 0.5 mg | Ozanimod 1 mg
Number analyzed (Participants) | 440 | 439 | 434
Participants
  Any TEAE | 365 | 326 | 324
  Any Moderate or Severe TEAE | 235 | 169 | 170
  Any Severe TEAE | 19 | 19 | 15
  Any Related TEAE | 30 | 12 | 19
  Any Serious TEAE | 28 | 31 | 28
  Any Related Serious TEAE | 0 | 1 | 1
  Any TEAE Leading to discontinuation of Study Drug | 18 | 14 | 13
  Any TEAE Leading to Study Withdrawal | 20 | 13 | 13
  Any Death on Study | 0 | 1 | 0

12. Post Hoc Outcome: Percent Change From Baseline in Normalized Brain Volume to Month 24 Based on Rank ANCOVA
Description: Brain volume (a measure of brain atrophy) was measured by brain MRI scans that were read at a centralized MRI reading facility by a blinded reader.
  Due to the non-normal distribution of the data for brain volume loss, the analyses for percent change from Baseline in normalized brain volume was repeated using rank-analysis of covariance (ANCOVA) and observed values.
Time Frame: Baseline and Month 24
Population: ITT Population; participants with available data at Baseline and Month 24
Measure: Median (Full Range); unit: percent change
Arm/Group | Interferon Beta-1a | Ozanimod 0.5 mg | Ozanimod 1 mg
Number analyzed (Participants) | 279 | 274 | 271
percent change | -0.940 [-5.33 to 1.44] | -0.710 [-5.21 to 1.36] | -0.690 [-5.65 to 0.85]
Statistical Analysis 1: Comparison: Interferon Beta-1a vs Ozanimod 1 mg; Test type: Superiority; p < 0.0001, Rank ANCOVA; Adjusted for region and Baseline EDSS category, with the dependent variable as the residual of the rank of brain volume at Baseline
Statistical Analysis 2: Comparison: Interferon Beta-1a vs Ozanimod 0.5 mg; Test type: Superiority; p < 0.0001, Rank ANCOVA; [statistical method as in outcome 12, analysis 1]

ADVERSE EVENTS:
Time Frame: From first dose of study drug to 28 days following the last dose of study drug; median duration of treatment was 24 months in each treatment group.
Description: The Safety Population included all participants who received at least 1 dose of study drug, analyzed according to the highest dose of ozanimod treatment actually received, not according to the treatment they were randomized to receive, if different.
Arm/Group | Interferon Beta-1a | Ozanimod 0.5 mg | Ozanimod 1 mg
All-Cause Mortality (participants affected / at risk) | 0/440 | 1/439 | 0/434
Serious Adverse Events (participants affected / at risk) | 28/440 | 31/439 | 28/434
Other Adverse Events (participants affected / at risk) | 275/440 | 185/439 | 199/434
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Interferon Beta-1a (N=440) | Ozanimod 0.5 mg (N=439) | Ozanimod 1 mg (N=434)
Acute Myocardial Infarction (Cardiac disorders) | 1 | 0 | 0
Atrial Fibrillation (Cardiac disorders) | 0 | 1 | 0
Sinus Tachycardia (Cardiac disorders) | 0 | 2 | 0
Supraventricular Tachycardia (Cardiac disorders) | 1 | 0 | 0
Goitre (Endocrine disorders) | 1 | 0 | 0
Keratoconus (Eye disorders) | 0 | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal Wall Haematoma (Gastrointestinal disorders) | 0 | 1 | 0
Large Intestine Polyp (Gastrointestinal disorders) | 1 | 0 | 0
Umbilical Hernia (Gastrointestinal disorders) | 0 | 0 | 1
Cyst (General disorders) | 0 | 1 | 0
Drowning (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 1
Cholecystitis Chronic (Hepatobiliary disorders) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 1 | 0
Hyperplastic Cholecystopathy (Hepatobiliary disorders) | 0 | 1 | 0
Acute Hepatitis B (Infections and infestations) | 0 | 1 | 0
Appendicitis (Infections and infestations) | 2 | 1 | 2
Chronic Sinusitis (Infections and infestations) | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 0
Pyelonephritis Acute (Infections and infestations) | 1 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 1
Ankle Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Carbon Monoxide Poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 1
Clavicle Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Comminuted Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Craniocerebral Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Intentional Overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0
Jaw Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Joint Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Ligament Sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Lower Limb Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Traumatic Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hepatic Enzyme Increased (Investigations) | 1 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Intervertebral Disc Disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Osteitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Chronic Lymphocytic Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Invasive Breast Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Malignant Melanoma In Situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Medulloblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Ovarian Fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Acoustic Neuritis (Nervous system disorders) | 0 | 0 | 1
Autonomic Nervous System Imbalance (Nervous system disorders) | 0 | 1 | 0
Central Nervous System Lesion (Nervous system disorders) | 0 | 0 | 1
Cerebral Haemorrhage (Nervous system disorders) | 0 | 0 | 1
Cerebral Infarction (Nervous system disorders) | 0 | 1 | 0
Cervical Radiculopathy (Nervous system disorders) | 0 | 1 | 0
Epilepsy (Nervous system disorders) | 1 | 1 | 1
Generalised Tonic-Clonic Seizure (Nervous system disorders) | 0 | 1 | 0
Guillain-Barre Syndrome (Nervous system disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 0
Lumbar Radiculopathy (Nervous system disorders) | 0 | 0 | 1
Multiple Sclerosis Relapse (Nervous system disorders) | 1 | 1 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 1
Sciatica (Nervous system disorders) | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 1 | 0
Speech Disorder (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0
Foetal Growth Restriction (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0
Placental Polyp (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1
Vanishing Twin Syndrome (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1
Suicide Attempt (Psychiatric disorders) | 0 | 1 | 0
Calculus Urinary (Renal and urinary disorders) | 0 | 0 | 1
Chronic Kidney Disease (Renal and urinary disorders) | 0 | 0 | 1
Renal Colic (Renal and urinary disorders) | 1 | 0 | 0
Urethral Stenosis (Renal and urinary disorders) | 0 | 0 | 1
Breast Cyst (Reproductive system and breast disorders) | 0 | 0 | 1
Cervical Polyp (Reproductive system and breast disorders) | 1 | 0 | 0
Dysfunctional Uterine Bleeding (Reproductive system and breast disorders) | 0 | 0 | 1
Endometriosis (Reproductive system and breast disorders) | 0 | 1 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 0 | 1
Ovarian Cyst (Reproductive system and breast disorders) | 0 | 0 | 2
Uterine Polyp (Reproductive system and breast disorders) | 1 | 0 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Skin Ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Interferon Beta-1a (N=440) | Ozanimod 0.5 mg (N=439) | Ozanimod 1 mg (N=434)
Influenza Like Illness (General disorders) | 215 | 26 | 27
Pyrexia (General disorders) | 27 | 12 | 10
Nasopharyngitis (Infections and infestations) | 48 | 59 | 68
Pharyngitis (Infections and infestations) | 15 | 24 | 17
Upper Respiratory Tract Infection (Infections and infestations) | 37 | 36 | 34
Urinary Tract Infection (Infections and infestations) | 17 | 22 | 19
Alanine Aminotransferase Increased (Investigations) | 20 | 29 | 26
Gamma-Glutamyltransferase Increased (Investigations) | 9 | 16 | 25
Headache (Nervous system disorders) | 53 | 55 | 44
Hypertension (Vascular disorders) | 14 | 20 | 24
Orthostatic Hypotension (Vascular disorders) | 27 | 27 | 30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results from a center cannot be submitted for publication before results of multicenter study are published unless it is more than one (1) year since study completion. Then, Investigator can publish if manuscript is submitted to Celgene sixty (60) days prior to submission. Investigator must delete confidential information before submission.

DOCUMENTS (2):
  • Study Protocol (2014-10-04): https://cdn.clinicaltrials.gov/large-docs/34/NCT02047734/Prot_000.pdf
  • Statistical Analysis Plan (2015-06-05): https://cdn.clinicaltrials.gov/large-docs/34/NCT02047734/SAP_001.pdf